CLINICAL TRIAL: NCT07284030
Title: The Effect of a Web-Based Supportive Psychoeducation Program on Psychological Well-Being, Quality of Life and Fear of Recurrence Applied to Patients Who Completed Active Breast Cancer Treatment
Brief Title: Psychoeducation and Well-Being After Breast Cancer
Acronym: Psychoeducatio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Nazli (Other)
Responsible Party: Sponsor-Investigator, Yasemin Nazli, Advanced Practice Nurse, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UskudarU 22.07.2024
Record Dates: First submitted 2025-12-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Cancer Survivors; Breast - Female; Psycho-Oncology
Keywords: Breast cancer; Psychoeducation; Web-based intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-arm parallel group randomized controlled trial comparing web-based psychoeducation program plus standard care versus standard care alone in breast cancer survivors.
Masking Description: This is an open-label study where masking is not feasible due to the nature of the intervention. Participants in the intervention group actively engage in weekly online psychoeducation sessions via Zoom and access the study website (www.onkodestek.org), while the control group receives standard care only. Both participants and researchers are aware of group allocation. The interactive nature of the psychoeducation program and direct participant-researcher contact during sessions make blinding impossible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive a 6-week web-based psychoeducation program plus standard care
  Interventions: Behavioral: Web-Based Psychoeducation Program
- Control Group (No Intervention): Participants receive standard care only

INTERVENTIONS:
Behavioral: Web-Based Psychoeducation Program — Six-week structured psychoeducation program delivered online through www.onkodestek.org website and weekly Zoom sessions. Topics include living with breast cancer, managing psychosocial issues, improving quality of life, psychological well-being, and finding hope and meaning. Each session lasts 30-45 minutes.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a web-based psychoeducation program on psychological well-being and quality of life in breast cancer survivors who completed active treatment at least one year earlier.

Seventy-two women will be randomly assigned to either a 6-week online psychoeducation program plus standard care or standard care alone. The intervention consists of weekly 30-45 minute online sessions focusing on coping strategies, psychosocial adjustment, quality of life, and psychological well-being.

Primary outcomes include psychological well-being, fear of cancer recurrence, quality of life, and hopelessness, assessed at baseline, post-intervention, and 2-month follow-up.

DETAILED DESCRIPTION:
This randomized controlled study investigates the effects of a structured web-based psychoeducation program on psychological outcomes in breast cancer survivors who have completed active treatment and are in remission for at least one year.

Eligible participants will be randomly allocated to an intervention group or a control group. The intervention group will receive a 6-week web-based psychoeducation program in addition to standard care, while the control group will receive standard care alone. The program is delivered through the online platform www.onkodestek.org and includes weekly live sessions conducted via Zoom, each lasting approximately 30-45 minutes.

The psychoeducation program addresses coping with breast cancer survivorship, psychosocial challenges, enhancement of psychological well-being, improvement of quality of life, and development of hope and meaning in life.

Psychological well-being, fear of cancer recurrence, quality of life, and hopelessness will be assessed at baseline, immediately after the intervention, and at 2-month follow-up using validated self-report measures. After study completion, participants in the control group will be granted access to the psychoeducation platform.

This study aims to assess whether web-based psychoeducation provides measurable psychological benefits for breast cancer survivors during the post-treatment survivorship period.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivors
* Completed active breast cancer treatment (surgery, chemotherapy, radiotherapy) at least 12 months ago
* Currently in remission (no evidence of active disease)
* Age between 18-65 years
* Able to read and write Turkish
* Access to computer or smartphone with internet connection
* Able to participate in online video sessions via Zoom
* Willing to provide informed consent

Exclusion Criteria:

* Current cancer recurrence or metastatic disease
* Active psychiatric disorder requiring treatment
* Cognitive impairment that prevents participation in online sessions
* Currently receiving active cancer treatment (excluding hormonal therapy)
* Participation in another psychosocial intervention study
* No internet access or inability to use web-based platforms
* Male breast cancer patients
* Unable to commit to 6-week program schedule

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Well-Being | Baseline, 6 weeks (post-intervention), and 2-month follow-up
  Measured by the Psychological Well-Being Scale
  Change in psychological well-being measured using the Psychological Well-Being Scale. The scale consists of 8 items rated on a 7-point Likert scale, with total scores ranging from 8 to 56. Higher scores indicate better psychological well-being.
Change in Fear of Cancer Recurrence | Baseline, 6 weeks (post-intervention), and 2-month follow-up
  Measured by the Fear of Cancer Recurrence Inventory
  Change in fear of cancer recurrence measured using the Fear of Cancer Recurrence Inventory. Items are scored on a 5-point Likert scale (0-4), with higher scores indicating greater fear of cancer recurrence.

SECONDARY OUTCOMES:
Change in Cancer-Related Quality of Life | Baseline, 6 weeks, and 2-month follow-up
  Measured by the EORTC QLQ-C30
  Change in cancer-related quality of life assessed using the EORTC QLQ-C30. Scores are transformed to a 0-100 scale. Higher scores indicate better quality of life for functional scales and global health status, and worse symptoms for symptom scales.
Change in Hopelessness | Baseline, 6 weeks, and 2-month follow-up
  Measured by the Beck Hopelessness Scale
  Change in hopelessness measured using the Beck Hopelessness Scale. The scale consists of 20 items with total scores ranging from 0 to 20. Higher scores indicate greater hopelessness.
Change in Breast Cancer-Specific Quality of Life | Baseline, 6 weeks, and 2-month follow-up
  Measured by the EORTC QLQ-BR23
  Change in breast cancer-specific quality of life measured using the EORTC QLQ-BR23. Scores are transformed to a 0-100 scale. Higher scores indicate better functioning and worse symptoms, depending on the subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Outpatient Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing decision is pending completion of the doctoral thesis and institutional review of data sharing policies. The decision will consider participant privacy, ethical requirements, and journal publication guidelines.

REFERENCES:
- [Background] Karsten MM, Roehle R, Albers S, Pross T, Hage AM, Weiler K, Fischer F, Rose M, Kuhn F, Blohmer JU. Real-world reference scores for EORTC QLQ-C30 and EORTC QLQ-BR23 in early breast cancer patients. Eur J Cancer. 2022 Mar;163:128-139. doi: 10.1016/j.ejca.2021.12.020. Epub 2022 Jan 20. PMID 35066338
- [Background] Mateu P, Teixidor-Batlle C, Suarez-Alcazar MP, Salas-Medina P, Catala-Vilaplana I, Hernando-Domingo C, Muriach M, Collado-Boira E. A qualitative case study of body image in women with breast cancer participating in an exercise program. Support Care Cancer. 2025 Oct 1;33(10):893. doi: 10.1007/s00520-025-09963-z. PMID 41032141